CLINICAL TRIAL: NCT03460964
Title: Evaluating Non-Invasive Measurement of Sweat Glucose of Patients With Diabetes - The ENGAGE Study
Brief Title: Measuring Sweat Glucose of Patients With Diabetes - The ENGAGE Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not perform accurate measures due to equipment and sensor issues.
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Edward Chao, Associate Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SD; UL1TR001442 (NIH)
Record Dates: First submitted 2018-02-23; First posted 2018-03-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus
Keywords: Sensor; Glucose; Sweat
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pilocarpine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Diabetes (Experimental): All participants will receive a minimum of 2 doses of pilocarpine 0.1 mL gel, applied to the skin via the glucose sensor to induce sweat. Glucose will be measured with both an adhesive (needle-free) glucose sensor and a glucometer, at fasting, and time points ranging from 15 to 200 minutes after consuming a standardized meal. There are no other interventions.
  Interventions: Device: Adhesive glucose sensor; Drug: Pilocarpine

INTERVENTIONS:
Device: Adhesive glucose sensor — Will assess sensor's performance by comparing readings from an adhesive glucose sensor with those from a glucometer.
  pilocarpine 0.1 mL gel, applied to the skin via the glucose sensor to induce sweat
Drug: Pilocarpine — Pilocarpine 0.1 mL gel, applied to the skin via the glucose sensor to induce sweat; will apply a minimum of 2 doses to each participant.

SUMMARY:
This pilot clinical trial will explore the accuracy and acceptability of a non-invasive, wearable glucose sensor in patients living with DM. This study will compare needleless glucose sensor readings from sweat with glucometer measurements from patients with any type of diabetes at fasting, and after a meal.

DETAILED DESCRIPTION:
There is an unmet need for a non-invasive glucose monitoring device. UCSD nanoengineers developed a flexible, ultra-thin sensor adherent to the skin, similar to a temporary tattoo. Sweat glucose correlates with blood glucose. This proposed study would be the first to examine this needle-free glucose sensor to measure glucose in endogenous sweat in individuals with DM, and would serve as the basis for future development of a continuous, non-invasive sensor. The investigators hypothesize that compared with a glucometer, a tattoo sensor can accurately measure sweat glucose in patients with DM.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with an existing diagnosis of diabetes mellitus, of any type, defined as having a fasting plasma glucose (FPG) > 126 mg/dL, or hemoglobin A1c (HbA1c) > 6.5%.
* Ability to provide informed consent for participation.

Exclusion Criteria:

* Individuals who do not have diabetes.
* Those who have an allergy to pilocarpine.
* Frequent episodes of low blood sugar (hypoglycemia), have no warning symptoms of hypoglycemia (hypoglycemia unawareness), or are at high risk of having hypoglycemia.
* If taking any of the following medications: any beta-blockers (including atenolol, carvedilol, metoprolol, and propanolol), chlorthalidone, hydrochlorothiazide, oxybutynin, and tiotropium.
* Individuals who have the following conditions, for which it is not safe to take pilocarpine, including:

Known or suspected gallstones or gallbladder disease

Kidney stones

Conditions that affect your thinking and/or memory, including Parkinson's disease and Alzheimer's disease

Asthma

Chronic obstructive pulmonary disease (COPD)

Glaucoma

Irritable Bowel Syndrome

Pregnancy - a pregnancy test will be obtained for each woman of child-bearing age.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Glucose measurements | Fasting, and time points ranging from 15 to 200 minutes after consuming a standardized meal. Participants can complete this study in 1 or 2 visits. The study team anticipates to complete this clinical trial in approximately 1 year.
  Comparing glucose readings from the sensor with those from a glucometer

SECONDARY OUTCOMES:
Acceptability of sensor | The investigators will collect this data at the completion of the study, after the fasting and post-meal glucose readings (at time points ranging from 15 to 200 minutes) are collected.
  Will ask participants for written and verbal feedback

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Chao, DO, Principal Investigator — UCSD
Locations (2):
- United States (2):
  - UCSD Altman Clinical and Translational Research Institute, San Diego, California
  - UCSD, San Diego, California

IPD SHARING:
Plan to Share IPD: Undecided